CLINICAL TRIAL: NCT02681393
Title: The Effectiveness of an Educational Brochure on Exercise and a Motivational Telephone Support in Physical Activity Maintenance for Stroke Survivors
Brief Title: Physical Activity Maintenance in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Ada Tang, Principal Investigator, McMaster University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PA Maintenance in Stroke
Record Dates: First submitted 2016-02-04; First posted 2016-02-12 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Stroke
Keywords: Physical activity, brochures, telephone support, stroke
MeSH Terms: conditions — Stroke; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brochure and Telephone Support (Experimental): Participants will receive both the Aerobic Exercise After Stroke educational brochure and 4 weekly motivational telephone support calls.
  Interventions: Behavioral: Brochure and Telephone Support
- Brochure Only (Active Comparator): Participants will receive the Aerobic Exercise After Stroke educational brochure only.
  Interventions: Behavioral: Brochure

INTERVENTIONS:
Behavioral: Brochure and Telephone Support — Participants will receive both the Aerobic Exercise After Stroke educational brochure and 4 weekly motivational telephone support calls.
  Arms: Brochure and Telephone Support
Behavioral: Brochure — Participants will receive both the Aerobic Exercise After Stroke educational brochure.
  Arms: Brochure Only

SUMMARY:
It is essential that individuals living with stroke engage in physical activity to improve cardiovascular risk factors and reduce the risk of stroke (Billinger et al, 2014). This objective of this study is to examine the effectiveness of an educational brochure that promotes exercise in people with stroke, combined with a motivational telephone support, on maintaining physical activity. Fifty participants with stroke will be enrolled. This study will provide insight into implementing effective tools that are designed to help individuals with stroke maintain physically active behaviours in the long-term.

DETAILED DESCRIPTION:
Study Design

This is a 4-week randomized controlled trial consisting of two groups: 1) participants who receive an educational brochure regarding physical activity after stroke, combined with motivational telephone support (intervention group), and 2) participants who receive the educational brochure alone (control group).

Interventions

Participants in the control group will be asked to devote approximately 30 minutes of their time to this study over the course of 4 weeks, and those in the intervention group will be involved for a total of 85 minutes.

1. Educational Brochure (both intervention and control groups): The educational brochure, Aerobic Exercise After Stroke, will be provided to all participants in the study. The brochure was created by researchers from the Canadian Partnership for Stroke Recovery and written for a stroke audience. It was designed to educate individuals with stroke about the benefits of aerobic exercise, exercise intensity, and provide a sample program.
2. Motivational Telephone Support (intervention group only): Motivational telephone support is an inexpensive way of supplementing the educational brochure for facilitating physical activity behaviors by establishing a personal connection and providing ongoing support and motivation. Participants in the intervention group will receive a total of 4 phone calls that will take place at 1-week intervals. Each telephone session will last approximately 15 minutes, where issues regarding ongoing physical activity, such as relapses and road blocks, will be addressed. Also, ongoing motivation and support will be provided as needed to re-direct participants back onto the path of physical activity engagement.

Statistical Analyses

Baseline participant characteristics will be analyzed using descriptive statistics. A two-way analysis on variance will be used to compare mean differences in physical activity and self-efficacy between the intervention and control group considering a group X time interaction

ELIGIBILITY:
Inclusion Criteria:

* Completed the intervention arm of a previous trial (Fit for Function)
* Living in the community
* Not involved in active rehabilitation

Exclusion Criteria:

* Musculoskeletal contraindications to exercise
* Unstable cardiovascular conditions
* Unstable medical conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Physical Activity | 4 weeks
  Rapid Assessment of Physical Activity questionnaire

SECONDARY OUTCOMES:
Physical Activity Self-Efficacy | 4 weeks
  General Self-Efficacy Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Ada Tang, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available.

REFERENCES:
- [Background] Billinger SA, Arena R, Bernhardt J, Eng JJ, Franklin BA, Johnson CM, MacKay-Lyons M, Macko RF, Mead GE, Roth EJ, Shaughnessy M, Tang A; American Heart Association Stroke Council; Council on Cardiovascular and Stroke Nursing; Council on Lifestyle and Cardiometabolic Health; Council on Epidemiology and Prevention; Council on Clinical Cardiology. Physical activity and exercise recommendations for stroke survivors: a statement for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2014 Aug;45(8):2532-53. doi: 10.1161/STR.0000000000000022. Epub 2014 May 20. PMID 24846875